CLINICAL TRIAL: NCT06960148
Title: Clinical Investigation of the Dentinal Hypersensitivity Reduction Efficacy of CSPR Toothpaste Containing 8% Arginine Compared to Colgate Cavity Protection Toothpaste Immediately Following Direct Topical Application of the Product and After Subsequent Brushing With the Product for Eight Weeks.
Brief Title: Dentinal Hypersensitivity Reduction Efficacy Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2025-02-SEN-CSPR-YPZ
Record Dates: First submitted 2025-04-22; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Sensitivity, Tooth
Keywords: hypersensitivity; dentin
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: This study will be monocentric, randomized, double-blind, two-treatment, parallel clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The tubes of test dentifrices will present the same shape/color to avoid that both investigators and subjects can identify the dentifrices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Toothpaste (Experimental): Subjects will be instructed to brush their teeth with their assigned teeth dentifrice and toothbrush twice daily
  Interventions: Drug: CSPR Toothpaste
- Control toothpaste (Active Comparator): Subjects will be instructed to brush their teeth with their assigned teeth dentifrice and toothbrush twice daily
  Interventions: Drug: Colgate Dental Cream Toothpaste

INTERVENTIONS:
Drug: CSPR Toothpaste — a commercially available 8% arginine toothpaste
  Arms: Test Toothpaste
Drug: Colgate Dental Cream Toothpaste — a commercially available fluoride toothpaste
  Arms: Control toothpaste

SUMMARY:
Assess the clinical efficacy of CSPR Toothpaste containing 8% arginine to provide dentinal hypersensitivity relief

DETAILED DESCRIPTION:
The objective of this study is to assess the clinical efficacy of CSPR Toothpaste containing 8% arginine to provide dentinal hypersensitivity relief (tactile and air blast) at instant, 3 days, 4 weeks and 8 weeks in comparison to Colgate Cavity Protection Toothpaste over an eight-week period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 18-70, inclusive.
* Availability for the eight-week duration of the study.
* Two sensitive teeth, which must be anterior to the molars, and demonstrate cervical erosion/abrasion or gingival recession.
* Qualifying response to tactile stimuli (Yeaple probe) as defined by a score between 10-50 gms. of force.
* Qualifying response to the air blast stimuli as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale.
* Subjects need to satisfy the qualifying response to stimuli for both the parameters assessed (tactile or air) on two teeth to be entered into the study.
* Good general health with no known allergies to products being tested.
* Use of a non-desensitizing dentifrice for three months prior to entry into the study.
* Signed Informed Consent Form.

Exclusion Criteria:

* Gross oral pathology, chronic disease, or history of allergy to test products. 2. Advanced periodontal disease or treatment for periodontal disease (including surgery) within the past twelve months.
* Sensitive teeth with a mobility greater than one.
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures.
* Current use of anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory drugs, or daily use of analgesics.
* Participation in a desensitizing dentifrice study or regular use of a desensitizing dentifrice within the past three months.
* Current participation in any other clinical study.
* Pregnant or lactating subjects.
* Allergies to oral care products, personal care consumer products, or their ingredients.
* Medical condition which prohibits not eating/drinking for 4 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Tactile Sensitivity using the Yeaple Electronic Force Sensing Probe | baseline, 3 day, 4 weeks, 8 weeks
  Tactile sensitivity will be assessed by use of Sensing Probe Yeaple Electronic Force Sensing Probe, Model 200A. Sensitivity will be defined by a score in the range of 10-50 gms. of force.
Air Sensitivity using the Schiff Cold Air Sensitivity Scale | baseline, 3 day, 4 weeks, 8 weeks
  The air will be directed at the exposed buccal surface of the sensitive tooth air delivered by a standard dental unit syringe at a measured temperature of 19-21°C (70°F[± 3°F].

CONTACTS AND LOCATIONS:
Locations (1):
- West China Dental Institute of Chengdu, Chengdu, Sichuan, China